CLINICAL TRIAL: NCT04900818
Title: A Phase 1 Study of TJ033721 in Subjects with Advanced or Metastatic Solid Tumors
Brief Title: Study of TJ033721 (givastomig) in Subjects with Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: I-Mab Biopharma US Limited (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TJ033721STM101
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor; Advanced Cancer; Metastatic Cancer; Gastric Cancer; Gastroesophageal Junction Carcinoma; Esophageal Adenocarcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Nivolumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TJ033721 (givastomig) (Experimental): Dose Escalation: TJ033721 will be administered at up to 8 dose levels (0.1, 0.3, 1, 3, 5, 8, 12 and 15 mg/kg) bi weekly (Q2W) and 1 dose level (18 mg/kg) every 3 weeks (Q3W)
  During dose expansion, TJ033721 will be administered Q2W, starting at the RP2D or MTD in dose escalation.
  Interventions: Drug: TJ033721 (givastomig)
- TJ033721 (givastomig) in combination with nivolumab and chemotherapy (Experimental): TJ033721 will be administered in combination with nivolumab and chemotherapy
  Interventions: Drug: TJ033721 (givastomig) , nivolumab, chemotherapy

INTERVENTIONS:
Drug: TJ033721 (givastomig) — Tetravalent IgG(H)-scFv fusion-type of bi-specific antibody (BsAb)
  Arms: TJ033721 (givastomig)
Drug: TJ033721 (givastomig) , nivolumab, chemotherapy — Tetravalent IgG(H)-scFv fusion-type of bi-specific antibody (BsAb), nivolumab, chemotherapy
  Arms: TJ033721 (givastomig) in combination with nivolumab and chemotherapy

SUMMARY:
This is an open label, multi-center, multiple dose Phase 1 study to evaluate the safety, tolerability, MTD PK, and PD of TJ033721 (givastomig) in subjects with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Part 1 - Monotherapy

• Subjects with advanced or metastatic solid tumor in subjects whose disease has progressed despite standard therapy, or who has no further standard therapy, or who is unsuitable for available standard treatment options.

Part 2 - Combination Therapy Subjects with treatment naïve locally advanced, unresectable or metastatic gastric, GEJ, esophageal adenocarcinoma;

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 with adequate organ function
* Have known PD-L1 status with prior testing by immunohistochemistry and a corresponding combined positive score (CPS)

For dose expansion and Part 2 Combination subjects:

• Must have CLDN18.2-positive tumor expression

Exclusion Criteria

* Prior exposure to CLDN18.2 -targeted therapy
* Prior exposure to 4-1BB agonists
* Second malignancy within the last 3 years with the exception of cutaneous squamous cell carcinoma or cutaneous basal cell carcinoma or cervical carcinoma in situ
* Known active or chronic Hepatitis B or Hepatitis C, other hepatitides
* Unstable/active ulcer or digestive tract bleeding within 6 weeks
* Active autoimmune disease requiring systemic treatment within the past 2 years
* Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment
* Known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment;
* New York Heart Association (NYHA) Class 3 or 4 congestive heart failure, severe/unstable angina, myocardial infarction (MI), symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack (TIA), arterial embolism, percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass grafting (CABG) in the previous 6 months
* Diagnosis of immunodeficiency such as known active HIV
* Any active infection requiring parenteral treatment

For Part 2 Combination subjects:

• Prior treatment with anti-PD-1 or PD-L1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | 28 days
Incidence and severity of AEs | Up to 100 days post last dose
  The CTCAE criteria will be used to assess adverse events on this trial.
Maximum tolerated or administered dose (MTD, MAD) | 28 Days
  Based on DLT definitions

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameters: AUC∞ | Up to 100 days post last dose
  Area under the curve from time zero extrapolated to infinity (AUC∞)
Pharmacokinetic (PK) Parameters: AUCt | up to 100 days post last dose
  AUC from time zero to the time of the last quantifiable concentration (AUC0-t)
Pharmacokinetic (PK) Parameters: Cmax | up to 100 days post last dose
  Maximum observed concentration
Pharmacokinetic Parameters: Tmax | up to 100 days post last dose
  Time of peak concentration (Tmax)
Pharmacokinetic Parameters: T1/2 | up to 100 days post last dose
  Investigational Product (IP) half-life (T1/2)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (11):
  - Stern Center for Cancer Clinical Trials and Research, Orange, California
  - UCHealth Cancer Care - Anschutz Medical Campus, Aurora, Colorado
  - Horizon Oncology Research, LLC., Layfayette, Indiana
  - Mass General Hospital, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - UW Carbone Cancer Center, Madison, Wisconsin
- China (10):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - HARBIN Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hongzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No